CLINICAL TRIAL: NCT00232635
Title: A Double-blind, Randomised, Placebo-controlled Study to Evaluate the Safety and Efficacy of A-60444 in Adults With RSV Infection Following Stem Cell Transplantation
Brief Title: A Study of the Safety and Efficacy of A-60444 in Adults With Respiratory Syncytial Virus (RSV) Infection Following HSCT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arrow Therapeutics (Industry)
Responsible Party: Arrow Therapeutics, Arrow Therapeutics
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CP204
Record Dates: First submitted 2005-10-04; First posted 2005-10-05 (Estimated); Last update posted 2010-02-12 (Estimated); Status verified 2010-02

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: RSV; HSCT; HEMATOPOIETIC STEM CELL TRANSPL
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: A-60444

SUMMARY:
Objectives

Primary Objectives:

* Pilot Study: A preliminary assessment of the exposure and safety of oral A-60444 in post-stem cell transplant patients with RSV infection.
* Main Study: To determine the antiviral effect of oral A-60444 versus placebo in post-stem cell transplant patients with RSV infection and to assess the safety of oral A-60444 in post-stem cell transplant patients with RSV infection.

Secondary Objectives:

* To study the pharmacokinetics of A-60444 in the presence of concomitant medications such as immunosuppressants and antifungals, in post-stem cell transplant patients with RSV infection.

Sample Size: Six patients will be included in the open, pilot phase of the study and there is an option to include a further 22 patients into the main, placebo-controlled study, depending on the pilot study findings. An independent Data Safety Monitoring Board will assess the findings of the pilot study.

DETAILED DESCRIPTION:
Clinical will be recorded daily. A-60444 PK will be studied pre-dose and at peak dose on the last day (Day 5) of dosing.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with RSV infection who have had a stem cell transplant.
2. Female patients must be of non-childbearing potential or have a negative pregnancy test prior to study start and be deemed not at risk of becoming pregnant. Females of non-childbearing potential are defined as women who have had a hysterectomy, bilateral oophorectomy, tubal ligation, or who have been post-menopausal for at least two years; or are considered to be sterile due to recent chemotherapy.
3. Aged between 18 and 65 years.
4. Patients who have given their written informed consent to participate in the study.
5. Patients who are willing and able to comply with the protocol and study procedures.

Exclusion Criteria:

1. Patients who have received an investigational drug within one month preceding the start of dosing.
2. Patients who have a documented history of allergy to benzodiazepines.
3. Patients with significant hepatic impairment (alanine transaminase [ALT] more than 5 x upper level of normal [ULN], total bilirubin more than 3 x ULN). Biochemistry data collected four weeks prior to screening is acceptable.
4. Patients, who in the opinion of their general practitioner or the Investigator, should not participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2005-09; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Reduction of viral load over time:
2-log reduction (by quantitative real time reverse transcription polymerase chain reaction [rtRT PCR]) in the RSV load of nasopharyngeal swabs in patients three days after treatment with A-60444, compared to patients treated with placebo

SECONDARY OUTCOMES:
Change in viral titre over treatment period
Safety, pharmacokinetics (PK)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen MacKinnon, Principal Investigator — Royal Free Hospital NHS Foundation Trust
Locations (1):
- Stephen MacKinnon, London, London, United Kingdom